CLINICAL TRIAL: NCT05241626
Title: Anterior Segment Optical Coherence Tomography Study of the Tear Film and Cornea in Thyroid Eye Diseases.
Brief Title: AS-OCT of the Cornea in Thyroid Diseases
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Salah, Dr Mohamed Salah, Minia University
Other Study IDs: 165-2021
Record Dates: First submitted 2022-02-04; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Thyroid Eye Disease
Keywords: Cornea- Tear film- AS-OCT
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1: 70 eyes of 35 patients of thyroid inactive disease
  Interventions: Diagnostic Test: AS-OCT
- Group 2: 70 eyes of 35 patients of thyroid active disease
  Interventions: Diagnostic Test: AS-OCT
- Group 3: Healthy controls
  Interventions: Diagnostic Test: AS-OCT

INTERVENTIONS:
Diagnostic Test: AS-OCT — Optical Coherence Tomography (OCT) creates detailed cross-sectional images of the anterior and posterior segments using low coherence interferometry. OCT is a noninvasive, real-time method for evaluating the tear meniscus, total corneal thickness (CT), and corneal epithelial thickness

SUMMARY:
use the anterior segment optical coherence tomography (AS-OCT) to evaluate the tear meniscus parameters, total corneal thickness (CT), and epithelial thickness in active and inactive thyroid eye diseases (TED) patients and compare them with age-matched controls.

DETAILED DESCRIPTION:
A prospective case-control clinical study. The study subjects were divided into 3 groups, group 1 of inactive thyroid patients, group 2 of active thyroid patients, and group 3 of healthy controls. The AS-OCT was used to measure lower tear meniscus parameters (tear meniscus height (TMH), tear meniscus depth (TMD), and tear meniscus area (TMA)), total CT and epithelial thickness

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were patients with thyroid disorders with age between 20 to 60 years with no ocular manifestations

Exclusion Criteria:

* being younger than 20 or older than 60, presence of systemic diseases as diabetes mellitus (DM) and autoimmune diseases as rheumatoid arthritis (RA) that may cause dry eye, previous ocular surgery, use of contact lenses, smokers, pregnant women, and breastfeeding women.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients were divided into 3 groups. Group 1 included 70 eyes of 35 patients of thyroid inactive disease, group 2 included 70 eyes of 35 patients of thyroid active disease, and group 3 included 70 eyes of 35 healthy controls
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-10-29 (Estimated); Study Completion 2022-10-29 (Estimated)

PRIMARY OUTCOMES:
Tear Meniscus Height | through study completion, an average of 6 months
  represented by a line joining the points corresponding to the upper corneo-meniscus junction to the lower eyelid-meniscus junction
Tear Meniscus Depth (TMD): | through study completion, an average of 6 months
  represented as the distance between the center of the upper boundary of the tear meniscus and the point at the bottom boundary where the cornea meets the eyelid
Tear Meniscus Area (TMA) | through study completion, an average of 6 months
  triangular area formed by the corneal anterior boundary, anterior boundary of the lower eyelid and anterior borderline of the tear meniscus

CONTACTS AND LOCATIONS:
Overall Officials: mohamed Mahmoud, Principal Investigator — Minia faculty of medicine
Locations (2):
- Egypt (2):
  - Minia Faculty of medicine, Minya
  - Minia University hospital, Minya

IPD SHARING:
Plan to Share IPD: No
IPD will not to be shared